CLINICAL TRIAL: NCT01098708
Title: Clinical Outcomes Validation in Non Ambulatory and Young Boys/Men With Duchenne Muscular Dystrophy (DMD)
Brief Title: This is a Study to Get More Information About Non Ambulatory Boys & Men With Duchenne Muscular Dystrophy
Acronym: DMD
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Nationwide Children's Hospital (Other); Boston Children's Hospital (Other); University of Minnesota (Other); University of California, Davis (Other)
Responsible Party: Principal Investigator, Anne Connolly, Professor of Neurology, Washington University School of Medicine
Other Study IDs: 10-0067
Record Dates: First submitted 2010-04-01; First posted 2010-04-05 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; non ambulatory
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Many therapeutic trials in DMD exclude non-ambulatory boys and men. Rate of progression in these non-ambulatory patients has been studied but consensus has not been reached for what measures are most reliable and reproducible. Furthermore, any treatment trial would be expected to demonstrate improved function and improvement in quality of life. Therefore, function, strength, and quality of life must be understood and standardized. While the goal of this proposal is to standardize clinical outcomes for therapeutic trials, careful understanding of the progression of DMD in non ambulatory boys may also lead to better medical treatment.

DETAILED DESCRIPTION:
For Non-ambulatory study, boys must be unable to walk without assistive devices for greater than or equal to one year.

Age at onset of study for non-ambulatory boys and men: greater than or equal to 7 years through age 22 years.

Genetic or biopsy confirmation of dystrophinopathy or clinical diagnosis of DMD with biopsy/genetic confirmation in a primary relative.

ELIGIBILITY:
Inclusion Criteria:

1. For Non-ambulatory study, boys must be unable to walk without assistive devices for greater than or equal to one year.
2. Age at onset of study for non-ambulatory boys and men: greater than or equal to 7 years through age 22 years.
3. Genetic or biopsy confirmation of dystrophinopathy or clinical diagnosis of DMD with biopsy/genetic confirmation in a primary relative.

Exclusion Criteria:

1. For Non-ambulatory study, the inability to understand and cooperate with the testing would exclude a subject. -

Ages: 7 Years to 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Non ambulatory boys and men with Duchenne muscular dystrophy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Dystrophin gene mutations that predispose to early onset cardiomyopathy | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anne Connolly, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No